CLINICAL TRIAL: NCT05521308
Title: Investigating Hearing Aid Frequency Response Curves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-3167
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: Hearing Loss; Hearing Aids; Frequency Response Curves
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss

STUDY DESIGN:
Intervention Model Description: The study is not a crossover study in it's true sense as there is only one arm. All participants will undergo all testing and will test each hearing aid variation. It should be noted that testing a different hearing aid variation (i.e., intervention) is done by simply clicking a button and having the hearing aid switch into a different variation. In this study, participants will go back and forth between different variations in order to make preference selections (Live Sound Quality task or US Matrix Test task).
  Additionally, in other outcome measures, participants will listen to pre-recorded stimuli that have the various frequency response curves applied. In this case, participants once again will be exposed to different hearing aid curves while simply listening via hearing aids and making preference selections. In the end, participants can be exposed to different hearing aid variations (i.e., interventions) simultaneously and also have the ability to go back and forth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Hearing Loss (Experimental): Individuals with hearing loss that meet the candidacy to wear hearing aids. All interventions are associated with the fitting of binaural hearing aids with various coupling methods. All participants will be assessed under all interventions.
  Interventions: Device: Hearing Aid - Standard Curve; Device: Hearing Aid - Variation #1; Device: Hearing Aid - Variation #2; Device: Hearing Aid - Variation #3; Device: Hearing Aid - Variation #4

INTERVENTIONS:
Device: Hearing Aid - Standard Curve — Our current hearing aids which will be programmed to our standard frequency response curve.
Device: Hearing Aid - Variation #1 — Hearing aids that will have the frequency response curve adjusted and fit to the participant's hearing loss.
Device: Hearing Aid - Variation #2 — Hearing aids that will have the frequency response curve adjusted and fit to the participant's hearing loss.
Device: Hearing Aid - Variation #3 — Hearing aids that will have the frequency response curve adjusted and fit to the participant's hearing loss.
Device: Hearing Aid - Variation #4 — Hearing aids that will have the frequency response curve adjusted and fit to the participant's hearing loss.

SUMMARY:
Internal research on the manufacturer's hearing aid products has idenitfied areas in which the investigators can improve the hearing aid frequency response curve. This study aims to investigate the current freqeuncy response curve in the manufacturer's products to variations of these curves to determine if hearing aid users prefer the variations over the manufacturer's standard curve.

DETAILED DESCRIPTION:
Internal testing has identified areas in which the investigators can improve the performance of the manufacturer's hearing aid products. This should potentially lead to increased hearing aid user satisfaction due to an improvement in sound quality. However, the investigators are currently unsure if implementing these new frequency response curves will be preferred by the manufacturer's clients. Therefore, a study is proposed in which hearing aid users will compare the manufacturer's current frequency response curve to variations made to the curve and determine which one they prefer while listening to live speech/music or while streaming speech/music.

ELIGIBILITY:
Inclusion Criteria:

* N2 - N4 Hearing losses
* Health Outer ear
* no visible congenital or traumatic deformity of the outer ear
* Symmetrical hearing loss - no air-bone gap greater than 10 dB at all 500, 1000, 2000, and 4000 Hz.
* Ability to answer questions and repeat sentences
* No history of problematic tinnitus or pain/discomfort from loud sounds
* No history of active drainage from the ears in the past 90 daysInformed consent as documented by signature
* Willingness to wear different styles of couplings
* Willingness to wear binaural fitting
* Experienced Users = more than 3 months of hearing aid experience. If not more than 3 months, they will be considered a new user (Experience will not exclude them from study, only will be used to categorize them)
* Ability to travel throughout facility

Exclusion Criteria:

* Contraindications to the medical device (MD) in this study (e.g. known hypersensitivity or allergy to the investigational products)
* Limited mobility/not able to come to the scheduled visit
* Inability to produce reliable hearing test results
* History of active drainage from the ear in the previous 90 days
* Abnormal appearance of the eardrum and ear canal.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Sonova - Kitchener, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaisberg J, Folkeard P, Levy S, Dundas D, Agrawal S, Scollie S. Sound Quality Ratings of Amplified Speech and Music Using a Direct Drive Hearing Aid: Effects of Bandwidth. Otol Neurotol. 2021 Feb 1;42(2):227-234. doi: 10.1097/MAO.0000000000002915. PMID 32976346
- [Background] Harianawala J, Galster J, Hornsby B. Psychometric Comparison of the Hearing in Noise Test and the American English Matrix Test. J Am Acad Audiol. 2019 Apr;30(4):315-326. doi: 10.3766/jaaa.17112. Epub 2018 Sep 25. PMID 30461418
- [Background] Wu YH, Stangl E, Chipara O, Hasan SS, Welhaven A, Oleson J. Characteristics of Real-World Signal to Noise Ratios and Speech Listening Situations of Older Adults With Mild to Moderate Hearing Loss. Ear Hear. 2018 Mar/Apr;39(2):293-304. doi: 10.1097/AUD.0000000000000486. PMID 29466265
- [Background] Neuman AC, Bakke MH, Hellman S, Levitt H. Effect of compression ratio in a slow-acting compression hearing aid: paired-comparison judgments of quality. J Acoust Soc Am. 1994 Sep;96(3):1471-8. doi: 10.1121/1.410289. PMID 7963011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted via an internal database. Participants were recruited from August 2022 - January 2023. Participants were mainly contacted via email or telephone and only seen at the listed study locations.
Pre-assignment Details: All participants were exposed to all interventions and as mentioned previously, participants were exposed to multiple interventions at once (i.e., different hearing aid freqeuncy response curves). All 33 participants completed each test (i.e., outcome measure) while exposed to all the interventions. Different periods represent the different outcome measures and in the order in which they occured are listed below. For the final analysis, results from 22 participants was used.
Period: US Matrix Test in Quiet - 30 Minutes
Arm/Group | Participants With Hearing Loss
Started | 33
Completed | 33 (4 participants data was used for piloting and subsequently removed for the final analysis. 5 participants data was ultimately removed due to hearing loss severity. 2 participants date was removed due to the inabiltiy to fully understand instructions or provide credible results. In the end, 22 participants data was used for the final data analysis.)
Not Completed | 0
Period: Sound Quality Ratings - Live - 1 Hour
Arm/Group | Participants With Hearing Loss
Started | 33
Completed | 33 (4 participants data was used for piloting and subsequently removed for the final analysis. 5 participants data was ultimately removed due to hearing loss severity. 2 participants date was removed due to the inabiltiy to fully understand instructions or provide credible results. In the end, 22 participants data was used for the final data analysis.)
Not Completed | 0
Period: Break Between Appointments 1 and 2
Arm/Group | Participants With Hearing Loss
Started | 33
Completed | 33
Not Completed | 0
Period: Streaming Sound Quality Ratings - 1 Hour
Arm/Group | Participants With Hearing Loss
Started | 33
Completed | 33 (4 participants data was used for piloting and subsequently removed for the final analysis. 5 participants data was ultimately removed due to hearing loss severity. 2 participants date was removed due to the inabiltiy to fully understand instructions or provide credible results. In the end, 22 participants data was used for the final data analysis.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 23
Age, Continuous [Mean (Full Range); unit: years] | 67.90 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 33
Hearing Thresholds - PTA (500,1000,2000,4000 Hz) [Mean (Full Range); unit: Decibals in Hearing Level (dB HL)] — Hearing thresholds are measured via a hearing test. A hearing test is conducted by a licensed professional who is trained to conduct hearing tests and determine the severity of a participant's hearing loss. Depending on the configuration and severity of the hearing loss dictates if participants meet the requirements to join a clinical study. Hearing thresholds are measured across various frequencies and certain frequencies can differ significantly between participants. The average of four frequencies (500, 1000, 2000, and 4000 Hz (i.e., Pure Tone Average (PTA)) summarizes a participants loss.
  Decibals in Hearing Level (dB HL) | 38.22 [25 to 52]

OUTCOME MEASURES:

1. Primary Outcome: Streaming Sound Quality Ratings
Description: Pre-filtered sound samples (based on frequency response curves) will be presented via a paired comparison task in which participants will determine which sound sample they prefer (i.e. better sound quality). Sound samples will be presented via hearing aids that are programmed to the participant's hearing loss.
  Participant's will be presented with two samples at a time and will choose which sample they prefer. For example, if Sample A was preferred over Sample B, then Sample A gets a score of 1. If Sample B was preferred over Sample A, then Sample B gets a score of 1. At the end of the task, scores will be tallied to determine which sample was preferred the most overall. There will be 5 different samples. The minimum value for the tallied score would be 0 (the sample was not preferred at all) and the maximum value would be 8 (implying that the sample was preferred in all trials). Higher scores mean that the sample was preferred more and lowers scores mean the sample was not preferred.
Time Frame: 60 minutes
Population: Out of 33 participants, 4 were pilot participants so their data was not analyzed for the final statistical analysis and 5 participants data was removed due to HL severity. Additionally, 2 participants data was removed for the final analysis as they struggled to understand the tasks within the study. In the end, 22 participants data was used for the final analysis.
Measure: Mean (Standard Error); unit: Mean Preference Counts per Participant
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 22
Mean Preference Counts per Participant
  Numbe of times Variation 1 was preferred over variation 2 across all genres per participant. | 10.7 (0.915)
  Numbe of times Variation 1 was preferred over variation 3 across all genres per participant. | 9.41 (0.805)
  Numbe of times Variation 2 was preferred over variation 1 across all genres per participant. | 7.46 (0.939)
  Number of times variation 2 was rated higher in sound quality than variation 3 across all samples | 5.91 (0.588)
  Numbe of times Variation 3 was preferred over variation 1 across all genres per participant. | 8.32 (0.815)
  Numbe of times Variation 3 was preferred over variation 2 across all genres per participant. | 8.05 (0.757)
  Numbe of times Variation 1 was rated the same as variation 2 across all genres per participant. | 3.13 (0.487)
  Numbe of times Variation 1 was rated the same as variation 3 across all genres per participant. | 3.59 (0.462)
  Numbe of times Variation 2 was rated the same as variation 3 across all genres per participant. | 6.73 (1.17)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; This is to see if there is a difference in preference count per participant between Variation #1, Variation #2 and Same counts; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.20 to 1.00]
Statistical Analysis 2: Comparison: Participants With Hearing Loss; This is to see if there is a difference between Variation #1 and Variation #2 preference counts per participant; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = 3.23, 95% CI 2-sided [0.41 to 6.05]
Statistical Analysis 3: Comparison: Participants With Hearing Loss; This is to see if there is a difference in preference count per participant between Variation #1, Variation #3 and Same counts; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [0.18 to 1.00]
Statistical Analysis 4: Comparison: Participants With Hearing Loss; This is to see if there is a difference between Variation #1 and Variation #3 preference counts per participant; Test type: Superiority; p = .54, t-test, 2 sided; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-1.36 to 3.55]
Statistical Analysis 5: Comparison: Participants With Hearing Loss; This is to see if there is a difference in preference count per participant between Variation #2, Variation #3, and Same counts; Test type: Superiority; p = .231, ANOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0 to 1.00]

2. Secondary Outcome: Sound Quality Rating - Live - Counts
Description: Participants will be asked to wear hearing aids and as they listen to speech in noise. They will be asked to toggle between two hearing aid programs and will be asked to make ratings in the lab and outdoors.
  Similar to Outcome 1, scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials run and samples tested). Higher scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Number; unit: Count of preferences
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 22
Count of preferences
  # of times the standard curve was rated higher in preference than variation 4 across samples - Lab | 79
  # of times the standard curve was rated lower in preference than variation 4 across samples - Lab | 95
  # of times the standard curve was rated the same as variation 4 in preference across samples - Lab | 46
  # of times the standard curve was rated higher in preference than variation4 across samples-Outdoors | 86
  # of times the standard curve was rated lower in preference than variation4 across samples-Outdoors | 104
  # of times the standard curve was rated the same as variation4 in preference across samples-Outdoors | 30

3. Secondary Outcome: Sound Quality Rating - Live - Preferences
Description: Participants will be asked to wear hearing aids and as they listen to speech in noise. They will be asked to toggle between two hearing aid programs and determine which program they prefer to listen to.
  Similar to Outcome 1, scores will be tallied at the end to see which program of the two was preferred more in the different listening environments. Scores can range from 0 (the program was not preferred at all) to unlimited (dependent on the numbers of trials run and samples tested). Highers scores will indicate that the program was preferred more than the other program and lowers scores mean the program was not preferred when compared to the other program.
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Number; unit: Count of preferences
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 22
Count of preferences
  # of participants that had an overall preference toward variation #4 vs. standard curve - Outdoors | 15
  # of participants that had an overall preference toward standard curve vs. Variation #4 - Outdoors | 6
  # of participants that had no preference toward standard curve vs. Variation #4 - Outdoors | 1
Statistical Analysis 1: Comparison: Participants With Hearing Loss; Test type: Superiority; p = .13, Chi-squared; This is to see if there is a difference in preference counts between standard curve, variation #4, and # of times they were rated as the same. -Indoor; Cramer's V = 0.14
Statistical Analysis 2: Comparison: Participants With Hearing Loss; Test type: Superiority; p = 0.04, Chi-squared — This is to see if there is a difference in preference counts between standard curve, variation #4, and # of time they were rated as the same. -Outdoor; Cramer's V = .20
Statistical Analysis 3: Comparison: Participants With Hearing Loss; The number of participants that showed overall preference toward variation #4 vs. the standard curve vs. no preference. - Outdoors; Test type: Superiority; p = 0.04, Chi-squared; Cramer's V = 0.2

4. Secondary Outcome: US Matrix Test in Quiet - SRT
Description: Oldenburg Sentence Test (OLSA) sentences were presented to participants while they were aided under the standard curve, aided under curve #4, and unaided. Participants are presented with sentences from a loudspeaker placed infront of them and asked to repeat what they heard. Correct repitition results in the next sentence to be presented at a lower sound level. Incorrect repetition results in an increase in presentation level for the next sentence. 20 sentences are presented for each conidition (i.e., unaided, aided with the standard curve, and aided under curve #4). Speech Recognition Threshold at 50% (SRT50) correctness scores were calculated and compared amongst the three conditions. SRT50 is measured in decibel (dB) which is a unit on scale. The scale has no upper or lower limits, however lower scores indicate better performance.
Time Frame: 30 Minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 22
decibels (dB)
  Unaided - Signal to Noise Ratio at 50% correct (SRT50) | 34.1 (9.9)
  Standard Curve - Signal to Noise Ratio at 50% correct (SRT50) | 25.8 (4.3)
  Variation 4 - Signal to Noise Ratio at 50% correct (SRT50) | 26.1 (4.21)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; Standard Curve vs Variation #4; Test type: Superiority; p < 0.001, ANOVA; Initally this is to see if there is a differnce between Unaided, Aided #1 and Aided #2; Effect Size = 0.26, 95% CI 2-sided [0.10 to 1.00]
Statistical Analysis 2: Comparison: Participants With Hearing Loss; Test type: Superiority; p = 0.855, t-test, 2 sided — Post-Hoc Pairwise Comparison; Standard Curve vs Variation #4; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-2.83 to 2.35]

ADVERSE EVENTS:
Time Frame: Participants were exposed to multiple interventions at once and had the ability to cycle through the various interventions (frequency curves). For this reason, adverse event data would have been collected per task and not intervention due to the quick exposure to multiple interventions. Adverse Event Data per participant was collected and is reported below. Sound Quality Ratings - Streaming - 60 minutes Sound Quality Ratings - Live - 60 minutes US Matrix Test Task in Quiet - 30 minutes
Arm/Group | Participants With Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT05521308/Prot_SAP_000.pdf